CLINICAL TRIAL: NCT04303767
Title: The Reparative Effect of Casein Phosphopeptide Amorphous Calcium Phosphate Varnish on Caries Affected Dentine in Primary Teeth (Randomized Controlled Clinical Trial)
Brief Title: The Effect of Casein Phosphopeptide Amorphous Calcium Phosphate on Affected Dentine
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00010556-IORG0008839
Record Dates: First submitted 2020-03-03; First posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Caries,Dental
Keywords: Casein Phosphopeptide Amorphous Calcium Phosphate; CPP-ACP; caries affected dentine; dentine repair; Atraumatic Restorative Treatment
MeSH Terms: conditions — Dental Caries | interventions — casein phosphopeptide-amorphous calcium phosphate nanocomplex; Dental Atraumatic Restorative Treatment

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test (ART + CPP-ACP) (Experimental): In this group, teeth selected will receive intervention with CPP-ACP and restorations with light cured Glass Ionomer restorations after excavating the carious lesions preserving the caries affected dentine using the ART
  Interventions: Drug: Casein phosphopeptide amorphous calcium phosphate; Procedure: Atraumatic restorative treatment
- Control (ART) (Active Comparator): in this group, teeth selected will receive restorations with light cured Glass Ionomer restorations after excavating the carious lesions preserving the caries affected dentine using the ART
  Interventions: Procedure: Atraumatic restorative treatment

INTERVENTIONS:
Drug: Casein phosphopeptide amorphous calcium phosphate — varnish containing calcium and phospate ions which act as a source for tooth remineralization
  Other Names: MI varnish
  Arms: Test (ART + CPP-ACP)
Procedure: Atraumatic restorative treatment — excavation of dental caries and restoring with light cured Glass Ionomer Restoration
  Other Names: ART

SUMMARY:
Teeth selected for intervention with Atraumatic Restorative Treatment will receive Glass Ionomer restorations (control) or MI varnish (test) before receiving the Glass Ionomer restoration

DETAILED DESCRIPTION:
Patients selected to participate in the study will be randomly assigned into 2 groups.

Group 1 (test): who will receive casein Phosphopeptide Amorphous Calcium Phosphate (CPP-ACP) + ART in the teeth selected, excavating only the caries infected dentine and preserving the caries affected dentine.

Group 2 (control): Who will receive ART only in the teeth selected, excavating only the caries infected dentine and preserving the caries affected dentine.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy patients.
2. Patients with an age range of 6-8 years old for clinical evaluation.
3. Patients ranking definitely positive or positive on Frankl scale.
4. Patients having at least 1 symptomless primary molar with caries extending to the dentine (International Caries Detection and Assessment System (ICDAS II) code 4, 5 & 6).
5. The presence of the permanent successors when examined by periapical X-ray.
6. Patients who will agree to participate in the study. For the ex-vivo sample

   1. Patients with an age range of 9-11 years old.
   2. The selected teeth should have more than half of their roots physiologically resorbed when examined by periapical X-ray.

Exclusion Criteria:

1. Patients with special health care needs (physical, mental or medical).
2. Primary molars that are mobile, ankylosed or have periapical pathology on initial examination clinically and radiographically.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 132 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the reparative ability of Casein Phosphopeptide Amorphous Calcium Phosphate varnish on caries affected dentine in primary molars. | 12 months
  this is by evaluating the clinical and radiographic data and also by descriptive histological assessment

OTHER OUTCOMES:
Evaluate and compare the clinical outcome of Atraumatic Restorative Treatment with and without Casein Phosphopeptide Amorphous Calcium Phosphate varnish placed on caries affected dentine in primary molars to evaluate the restoration success or failure. | 12 months
  clinical criteria and ART success criteria will be assessed
Assess the radiographic success of Atraumatic Restorative Treatment with and without CPP-ACP varnish placed on caries affected dentine in primary molars by measuring the grey value radiographically using Image J software. | 12 months
  radiographic success of the teeth and radiographic density measures will be assessed
Assess histologically the quality of the formed dentine using the Polarized Light Microscope and Scanning Electron Microscope. | throughout the 12 months
  polarized light microscope and scanning electron microscope will be used to describe the repaired dentine and the bacterial load

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A. Bayoumi, MSc, Principal Investigator — Pharos University in Alexandria; Azza G. Hanno, Professor, Study Director — Alexandria University; Karin M. Dowidar, Professor, Study Director — Alexandria University; Samia S. Omar, Professor, Study Director — Alexandria University
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt